CLINICAL TRIAL: NCT03895320
Title: Protecting Our Future: Promotion of Protective Sexual Health Practices Among Native American Youth and Young Adults Through an Assets-based Self-care Intervention
Brief Title: Protecting Our Future Generation: Promotion of Protective Sexual Health Practices Among Native American Youth and Young Adults Through an Assets-based Self-care Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Native American Research Center for Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 8964; IRB00008964 (Other: JHSPH IRB)
Record Dates: First submitted 2019-03-15; First posted 2019-03-29 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Sexual Behavior; Unprotected Sex; Gonorrhea; Chlamydia; Trichomonas; Sexually Transmitted Diseases; Adolescent Behavior; Self Evaluation
Keywords: Native American; Youth; Young Adults; STI Screening; Self Administered Sample Collection
MeSH Terms: conditions — Sexual Behavior; Unsafe Sex; Gonorrhea; Chlamydia Infections; Trichomonas Infections; Sexually Transmitted Diseases; Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Program (Experimental): The intervention and control programs will consist of similar, but not identical components. The intervention will include a) a brief self-assessment (also called 'quiz'), b) score, and c) personalized messaging. For the intervention program, the self-assessment ('Sexual Health Quiz'), score ('Sexual Health Score') and messaging ('Sexual Health Messaging') will pertain to sexual and reproductive health. For the intervention program, the self-assessment, will include a valid clinical prediction tool, established to predict STI positivity. Short messages that indicate key steps the person can take to lower their risk for STIs will be displayed on the screen after the risk score. The program will be delivered via tablet. All participants regardless of randomization group, will be offered a STI screening kit immediately after receipt of their respective program.
  Interventions: Behavioral: Sexual Health Risk Assessment; Behavioral: Sexual Health Score; Behavioral: Sexual Health Messaging; Behavioral: STI Screening
- Control Program (Other): The intervention and control programs will consist of similar, but not identical components. The Control Program will include a) a brief self-assessment (also called 'quiz'), b) score, and c) personalized messaging. For the Control Program, the self-assessment ('Water Sugar Sweetened Beverages (SSB) Quiz'), score ('Water SSB Score') and messaging ('Water SSB Messaging') will pertain to consumption of water, soda and sugar sweetened beverages. There will not be a comparable clinical prediction tool in the control self-assessment. However, based on the answers given on the control quiz, steps the control participant can take to meet the recommended daily intake of water and sugar sweetened beverages will be displayed on the screen after they complete the quiz. The control program will be delivered via tablet. All participants regardless of randomization group, will be offered a STI screening kit immediately after receipt of their respective program.
  Interventions: Behavioral: Water SSB Quiz; Behavioral: Water SSB Score; Behavioral: Water SSB Messaging; Behavioral: STI Screening

INTERVENTIONS:
Behavioral: Sexual Health Risk Assessment — The self-assessment ('Sexual Health Risk Assessment'), will pertain to sexual and reproductive health. The self-assessment, will include a valid clinical prediction tool, established to predict STI positivity.
  Arms: Intervention Program
Behavioral: Sexual Health Score — The results of the 'Sexual Health Risk Assessment' will produce a score ('Sexual Health Score'). The 'Sexual Health Score' will be presented as a number (0/10) and will be organized by category: Low, Medium or High Risk.
  Arms: Intervention Program
Behavioral: Sexual Health Messaging — After the score ('Sexual Health Score') the participant will receive personalized messaging ('Sexual Health Messaging') that relates to their score and risk level (i.e. Low, Medium or High). Short messages that indicate key steps the person can take to lower their risk for STIs will be displayed on the screen that correspond to their 'Sexual Health Score.'
  Arms: Intervention Program
Behavioral: Water SSB Quiz — The self-assessment ('Water SSB Quiz') will pertain to consumption of water, soda and sugar sweetened beverages. There will not be a comparable clinical prediction tool in the control self-assessment ('Water SSB Quiz).
  Arms: Control Program
Behavioral: Water SSB Score — The results of the 'Water SSB Quiz' will produce a score ('Water SSB Score'). The 'Water SSB Score' will be presented as a number (0/10).
  Arms: Control Program
Behavioral: Water SSB Messaging — After the score ('Water SSB Score') the participant will receive personalized messaging ('Water SSB Messaging') that relates to their score. Short messages that indicate key steps the person can take to meet the recommended daily intake for water and sugar sweetened beverages will be displayed on the screen that correspond to their 'Water SSB Score.'
  Arms: Control Program
Behavioral: STI Screening — All participants regardless of group, will be offered a STI screening kit immediately after receipt of their respective program (intervention or control). Participants will have the option of completing the kit at the first study visit, taking it with them after the first study visit is over, or receiving it later from one of our staff either at our local project office or the kit can be dropped off at a location the participant chooses. Completed kits can be returned to our office or picked up by a study staff. (NOTE: while the STI screening kit will be available to all participants should they request it at subsequent study visits, e.g. the 3- and 6-month follow-ups, the STI screening kit will only be explicitly offered by the study team at the first study visit immediately after participants complete their respective quiz).

SUMMARY:
The aim of this research protocol is to test the efficacy of a self-care intervention through a randomized controlled trial (RCT), for increasing protective sexual health behaviors among youth in the participating Native American community. The investigators will randomize 450 youth and young adults ages 14-26 to the self-care intervention or a control program. Efficacy data will be collected up to 6 months post-intervention. The primary outcome will be uptake of sexually transmitted infection (STI) screening. Secondary outcomes will include: a) sexual risk and protective behaviors; and b) psychosocial assets and resources. The investigators hypothesize the self-care intervention will increase protective behaviors by: i) helping youth gain knowledge of their own sexual health risks, assets and resources; ii) motivating protection of those assets and resources; and iii) encouraging good health practices and making responsible choices.

DETAILED DESCRIPTION:
The proposed study is a RCT to test the efficacy of a self-care intervention for sexual health promotion among youth and young adults in a participating Native American community. The goal of the intervention is to increase protective sexual health practices. The investigators will compare outcomes between two groups: the 1) experimental group and the 2) comparison group. Youth will be enrolled in the study and assessed at baseline, 3-months and 6-months post-intervention. Participants ages 14-26 will be enrolled through a non-probability sampling frame at: a) the local Indian Health Service (IHS) facility, including the Emergency Department waiting room; b) local schools; c) during health fairs and other community-based events; and d) other community gathering spots. Eligible individuals will be of Native American ethnicity, 14-26 years of age, and have primary residence and/or employment within the participating tribe's reservation. Research staff will screen potential participants for inclusion/exclusion criteria, explain study goals and procedures, and administer informed consent. After obtaining participant consent, participants will complete a baseline assessment and then be randomized to receive the self-care intervention or a control program. Follow-up assessments will be administered at 3-months and 6-months post-intervention for all study participants. Each assessment is expected to take 20-30 minutes to complete. The baseline assessment will take place at the location of recruitment and consent; follow-up assessments will take place at home or in a private location. All assessments will be self-administered on tablets using REDCap mobile technology.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-26
2. Native American ethnicity
3. Membership in the participating Native American community. (Study participation is open to all Native American individuals who live on the participating Tribe's Reservation, on/near the border, and/or are employed on the participating Tribe's Reservation).
4. Have had sex at least once in their lifetime (vaginal)
5. Participant must have their own cell phone and agree to receiving generic text messages and phone calls from study staff
6. All participants must sign informed consent

Exclusion Criteria:

1. Unwilling to be randomized
2. Inability to participate in full intervention or evaluation (e.g., planned move, residential treatment, etc.)

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 219 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in self-reported STI screening at 3-months and 6-months | 3-months and 6-months
  Difference in completion of self-administered screening kit for gonorrhea, chlamydia, and trichomonas between intervention and control groups at 3-months and 6-months. Participants report if they completed a self-administered test at each time point.

SECONDARY OUTCOMES:
Sex without condom | 3-months and 6-months
  Change in sex without a condom, between intervention and control groups at 3-months and 6-months, as measured by a self-report questionnaire. A dichotomous scale will be used (0, No; 1, Yes). A higher value indicates a worse outcome.
Sex without birth control | 3-months and 6-months
  Change in sex without birth control, between intervention and control groups at 3-months and 6-months, as measured by a self-report questionnaire. A dichotomous scale will be used (0, No; 1, Yes). A higher value indicates a worse outcome.
Multiple partners | 3-months and 6-months
  Change in number of sexual partners, between intervention and control groups at 3-months and 6-months, as measured by a self-report questionnaire. A dichotomous scale will be used (0, No; 1, Yes). A higher value indicates a worse outcome.
New partners | 3-months and 6-months
  Change in number of new sexual partners, between intervention and control groups at 3-months and 6-months, as measured by a self-report questionnaire. A dichotomous scale will be used (0, No; 1, Yes). A higher value indicates a worse outcome.
Concurrent partners | 3-months and 6-months
  Change in number of new sexual partners, between intervention and control groups at 3-months and 6-months, as measured by a self-report questionnaire. A dichotomous scale will be used (0, No; 1, Yes). A higher value indicates a worse outcome.
Current symptoms of STI | 3-months and 6-months
  Change in current symptoms of STI, between intervention and control groups at 3-months and 6-months, as measured by a self-report questionnaire. A dichotomous scale will be used (0, No; 1, Yes). A higher value indicates a worse outcome.
Alcohol and drug use | 3-months and 6-months
  Change in frequency of alcohol and drug use, between intervention and control groups at 3-months and 6-months, as measured by a self-report questionnaire. A dichotomous scale will be used (0, No; 1, Yes). A higher value indicates a worse outcome.
Alcohol and drug use before sex | 3-months and 6-months
  Change in frequency of alcohol and drug use before sex, between intervention and control groups at 3-months and 6-months, as measured by a self-report questionnaire. A dichotomous scale will be used (0, No; 1, Yes). A higher value indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Francene Larzelere, D BH, Study Director — Johns Hopkins Bloomberg School of Public Health; Rachel Chambers, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for American Indian Health, Whiteriver, Arizona, United States

REFERENCES:
- [Derived] Lauren T, Catherine S, Rachel C, Hima P, Angelita L, Shauntel L, Laura M, Anna S, Anne R, Mariddie C, Charlotte G. Protecting our future generation: study protocol for a randomized controlled trial evaluating a sexual health self-care intervention with Native American youth and young adults. BMC Public Health. 2019 Dec 2;19(1):1614. doi: 10.1186/s12889-019-7956-x. PMID 31791323